CLINICAL TRIAL: NCT02014610
Title: Leukocyte Counts and Initial Presentation of Cardiovascular Diseases: a CALIBER Study
Brief Title: White Blood Cell Counts and Onset of Cardiovascular Diseases: a CALIBER Study
Acronym: CALIBER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University College, London (Other)
Collaborators: Wellcome Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Medical Research Council (Other Government); London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: CALIBER 13-15; 0938/30/Z/10/Z (Other Grant/Funding Number: Wellcome Trust); RP-PG-0407-10314 (Other Grant/Funding Number: UK National Institute for Health Research); 086091/Z/08/Z (Other Grant/Funding Number: Wellcome Trust)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Abdominal Aortic Aneurysm; Coronary Artery Disease; Stroke; Heart Failure; Peripheral Arterial Disease
Keywords: Neutrophil; Lymphocyte; Eosinophil; Leukocyte count; Cardiovascular disease; Atherosclerosis; Monocyte; Basophil
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Coronary Artery Disease; Stroke; Heart Failure; Peripheral Arterial Disease; Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The complete blood count is a commonly performed blood test, and previous small studies have suggested that the counts of some types of white blood cell in the complete blood count may be related to the onset of cardiovascular diseases such as stroke and heart attack. This is of interest because this information may help to predict strokes or heart attacks and may guide new therapies which act on white blood cells to reduce the risk of cardiovascular disease.

The hypothesis is that counts of particular types of white blood cell are associated with a range of cardiovascular diseases.

DETAILED DESCRIPTION:
There is evidence from epidemiological studies that counts of some types of white blood cell, such as neutrophils, are associated with increased incidence of coronary disease. Associations with other initial presentations of cardiovascular diseases have not been studied in large cohorts, but may be of interest for use in risk prediction or to guide therapeutic strategies.

The aim of this study is to estimate associations between counts of lymphocytes, neutrophils, eosinophils, monocytes and basophils, and initial presentation of a range of cardiovascular diseases.

The study will use data from the CALIBER dataset of clinically collected electronic health record data from England. Patients enter the study when they have a full blood count (complete blood count) recorded in the dataset, and they are followed up until they experience one of the cardiovascular endpoints, death or transfer out of the participating primary care practice.

This study is part of the CALIBER (Cardiovascular disease research using linked bespoke studies and electronic records) programme funded over 5 years from the National Institute for Health Research (NIHR) and Wellcome Trust. The central theme of the CALIBER research is linkage of the Myocardial Ischaemia National Audit Project (MINAP) with primary care (Clinical Practice Research Datalink) and other resources. The overarching aim of CALIBER is to better understand the aetiology and prognosis of specific coronary phenotypes across a range of causal domains, particularly where electronic records provide a contribution beyond traditional studies. CALIBER has received both Ethics approval (ref 09/H0810/16) and ECC approval (ref ECC 2-06(b)/2009 CALIBER dataset).

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 30 and over, registered with a participating general practice during the study period.

Exclusion Criteria:

* Patients without a measurement of full blood count during the study period.
* Patients with prior atherosclerotic disease, as recorded in primary care or hospitalisation data.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Cohort study of patients in the CALIBER database who have a record of a full blood count (complete blood count) during the study period while registered at one of 225 general practices contributing data to CPRD (the Clinical Practice Research Datalink) and consenting to data linkage.
Sampling Method: Non-Probability Sample
Enrollment: 800000 (Estimated)
Dates: Start 1997-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Initial presentation of cardiovascular disease | 10 years
  First recorded diagnosis of cardiovascular disease during follow-up: ventricular arrhythmia / sudden cardiac death, heart failure, unheralded coronary death, myocardial infarction, unstable angina, stable angina, abdominal aortic aneurysm, peripheral arterial disease, subarachnoid haemorrhage, intracerebral haemorrhage, ischaemic stroke, transient ischaemic attack

SECONDARY OUTCOMES:
All cause mortality | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Anoop D Shah, MRCP, Principal Investigator — University College, London; Harry Hemingway, FRCP, Study Director — University College, London

REFERENCES:
- [Background] Denaxas SC, George J, Herrett E, Shah AD, Kalra D, Hingorani AD, Kivimaki M, Timmis AD, Smeeth L, Hemingway H. Data resource profile: cardiovascular disease research using linked bespoke studies and electronic health records (CALIBER). Int J Epidemiol. 2012 Dec;41(6):1625-38. doi: 10.1093/ije/dys188. Epub 2012 Dec 5. PMID 23220717
- [Derived] Shah AD, Denaxas S, Nicholas O, Hingorani AD, Hemingway H. Neutrophil Counts and Initial Presentation of 12 Cardiovascular Diseases: A CALIBER Cohort Study. J Am Coll Cardiol. 2017 Mar 7;69(9):1160-1169. doi: 10.1016/j.jacc.2016.12.022. PMID 28254179
- [Derived] Shah AD, Thornley S, Chung SC, Denaxas S, Jackson R, Hemingway H. White cell count in the normal range and short-term and long-term mortality: international comparisons of electronic health record cohorts in England and New Zealand. BMJ Open. 2017 Feb 17;7(2):e013100. doi: 10.1136/bmjopen-2016-013100. PMID 28213596
- [Derived] Shah AD, Denaxas S, Nicholas O, Hingorani AD, Hemingway H. Low eosinophil and low lymphocyte counts and the incidence of 12 cardiovascular diseases: a CALIBER cohort study. Open Heart. 2016 Sep 5;3(2):e000477. doi: 10.1136/openhrt-2016-000477. eCollection 2016. PMID 27621833
- See also: CALIBER web site and data portal — https://www.caliberresearch.org/